CLINICAL TRIAL: NCT04948788
Title: A Phase I/ II Study of SHR1459 in Combination With YY-20394 in Recurrent and Refractory B-cell Non-Hodgkin's Lymphoma in Adults
Brief Title: SHR1459 in Combination With YY-20394 in Recurrent and Refractory B-cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR1459-II-201
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-06

CONDITIONS: Recurrent and Refractory B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — gemcitabine-oxaliplatin regimen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR1459 + YY-20394 (Stage 1) (Experimental)
  Interventions: Drug: SHR1459 ；YY-20394
- SHR1459 + YY-20394 (Stage 2) (Experimental)
  Interventions: Drug: SHR1459 ；YY-20394
- GemOx (Stage 2) (Experimental)
  Interventions: Drug: Gemcitabine-Oxaliplatin

INTERVENTIONS:
Drug: SHR1459 ；YY-20394 — SHR1459 plus YY-20394
  Arms: SHR1459 + YY-20394 (Stage 1)
Drug: SHR1459 ；YY-20394 — SHR1459 plus YY-20394
  Arms: SHR1459 + YY-20394 (Stage 2)
Drug: Gemcitabine-Oxaliplatin — Gemcitabine-Oxaliplatin
  Arms: GemOx (Stage 2)

SUMMARY:
The study is evaluating the efficacy, and safety of SHR1459 combined with YY-20394 for Recurrent and refractory B-cell non-Hodgkin's lymphoma in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of B-cell NHL such as DLBCL, FL and MCL
2. Patients received at least 2 lines of systemic therapy
3. Previously received anti- CD20 treatment
4. Patients in stage II should also be unsuitable or unwilling to receive allogeneic hematopoietic stem cell transplantation
5. Patients must have an acceptable organ function

Exclusion Criteria:

1. Previously treated with PI3K inhibitors or BTK inhibitors
2. Unresolved toxicity of CTCAE grade > 1 from prior anti-lymphoma therapy
3. Chemotherapy or other investigational therapy within 28 days (or 5 times the half-life time, whichever is shorter) before starting cycle 1
4. Significant concurrent medical disease or condition which according to the investigators' judgement
5. Active hepatitis B, C or HIV infection
6. Infection requiring treatment 2 weeks prior to the first dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Stage 1: MTD （Maximum tolerated dose）or RP2D（Recommended Phase II Dose) of SHR1459 and YY-20394; | Minimum observation period is 28 days for the maximum dose cohort
Stage 2: Overall response rate (ORR) | 8 weeks after last patient first visit (LPFV)

SECONDARY OUTCOMES:
Incidence of Adverse Events | At every treatment and follow up visit until disease progression. Expected to be for up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality, China